CLINICAL TRIAL: NCT06945757
Title: Evaluation of an Oncological Rehabilitation Program as Part of the Promotion of Therapeutic Physical Activity in Adults Cancer Patients
Acronym: OnkoREHAB
Status: Recruiting | Type: Observational
Sponsor: Andrea Fontana (Other)
Responsible Party: Sponsor-Investigator, Andrea Fontana, Dr. med. Andrea Fontana, MSc, PhD, Principal Investigator, Luzerner Kantonsspital
Organization: Luzerner Kantonsspital (Other)
Other Study IDs: OnkoREHAB
Record Dates: First submitted 2025-01-08; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Cancer Rehabilitation
Keywords: Cancer; physical activity; rehabilitation
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients starting, undergoing or having completed chemotherapy
  Interventions: Other: Physical Exercise

INTERVENTIONS:
Other: Physical Exercise — Patients will participate in the routine rehabilitation program for 12 weeks, consisting of two 1h30 one-to-one sessions per week of physical activity administered by experienced physical therapist. Both sessions of the week are tailored to the need of the individual participant and are typically structured as follow:
  * 10 minutes of warming up by light exercises
  * 20 minutes of coordination exercises
  * 20 minutes of strengths exercises
  * 20 minutes of mobility exercises
  * 10-15 minutes of cool down and stretching
  Patients will further benefit during the 12-weeks program of several individual encounters with a psycho-oncologist, a nurse specialized in cognitive support and a nutritionist. Furthermore, a dietician will conduct an introductory evaluation, several intermediate evaluations and a final evaluation on nutritional status and habits of the patients.

SUMMARY:
It is estimated that there were 19.3 million newly diagnosed cancer cases and almost 10 million cancer-related deaths globally in 2020. Despite the numerous advances in cancer treatment, cancer incidence and mortality have been increasing over the years, thus making cancer one of the greatest health threats to human beings.

In recent decades, the advent of novel therapies in cancer has significantly prolonged the survival of oncological patients, yet many of these individuals are left with residual deﬁcits, particularly motor and neurological, as well as cancer-related fatigue and depression.

Exercise-based cancer rehabilitation is one of the main strategies which has been proved to be an effective way to improve the quality of life of cancer survivors. There are three main types of exercise training included as part of cancer rehabilitation: resistance exercise, aerobic exercise, and the combination of both. Furthermore, cognitive, and psychological support during this period might have a synergistic effect with physical activity.

Although rehabilitation procedures are very well established after cardiovascular and neurological events, such as myocardial infarction or stroke, their role in oncology has only marginally been investigated nor completely accepted by the medical community. Nevertheless, cumulating evidence with clinical experience suggests that physical activity has emerged as an important complementary supportive care for cancer patients and can improve the care of patients with cancer and their quality of life.

General clinical guidelines recommend that cancer rehabilitation begins ideally at the time of cancer diagnosis and continues through and beyond cancer treatment, but this is rarely done in clinical practice.There has been an effort to conduct qualitative studies to evaluate the effects of physical activity on cancer patients, with a particular focus on factors influencing an active lifestyle in cancer patients during or right after conclusion of oncological treatments. Most of these studies have been regrouping patients with a specific cancer type, with a particular focus on breast cancer. Nevertheless, it is relatively difficult to gain evidence from single qualitative studies on it owns, mostly due to the variety of qualitative methodologies employed and the lack of consistent results.

The principal aim of cancer rehabilitation is to help patients regain functioning, promote their independence and to increase their social participation, no matter how long or short the timescale. To evaluate and optimize rehabilitation, it is therefore very important to measure its outcomes in a structured and reproducible way. In recent exercise guidelines, most of the available evidence on the efficacy of oncology rehabilitation is derived from randomized controlled trials (RCTs), which have strengthened the body of proof for the efficacy of exercise in cancer rehabilitation, but on the other side they have been reported to lack generalizability to the clinical setting. In these trials, patients often must meet pre-specified criteria (e.g., diagnosis, disease stage, age) to be eligible for enrolment in RCTs and must give consent to participate. This might bias results toward a healthier, fitter, and more motivated population, which may not be comparable to a broader population of cancer survivors. While RCTs have the most powerful study design to investigate the efficacy of rehabilitation in a specific population under ideal circumstances, observational studies may be more appropriate to evaluate interventions in daily practice and in more heterogeneous populations with complex, chronic diseases such as cancer.

A major determinant of functional capacity is exercise behaviour. The beneficial effects of physical exercise have been shown to improve multiple aspects of health in cancer survivors, including quality of life, fatigue, as well as all cause and cancer specific mortality.

Physical impairments and psychosocial symptoms should be assessed and treated concomitantly, and lifestyle and exercise interventions provided to optimize functioning and quality of life (QoL). Quality of life can be defined as a multidimensional structure that reﬂects a person's subjective evaluation of their well-being and functioning across multiple life domains, and each of these should be specifically addressed by cancer support services. According to Ferrans, five dimensions of QoL have been described: physical; functional; psychological/emotional; social; and spiritual. Ideally, all these dimensions should be explored in cancer patients in relation to exercise.

Metanalysis across several studies have shown that patients noticed consistent improvements in their physical and psychological functioning and health. Furthermore, many patients have reported that exercise has helped them to better manage the physical consequences of cancer and its treatment, contributing to their overall fitness.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the feasibility, acceptability, and effectiveness of a 12-weeks rehabilitation program on cancer patients currently undergoing or having just completed any type of oncological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, with an history of malignancy, who are going to start, are currently undergoing primary cancer treatment or just ended their oncological treatment, independent of cancer type.
* Age between 18 and 80 years.
* Available 2 days per week all along the program duration.

Exclusion Criteria:

* Major foreseeable risk of impossibility to participate in the session due to therapeutic toxicities or other reasons that may lead to a sustainable lack of compliance incompatible with the continuation of the program.
* Patients not having a full decisional capacity
* Patients not able to maintain a satisfactory professional or personal aptitude during the program.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncological Patients
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy | 36 months
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire designed to measure quality of life. The FACT-G measures five domains of quality of life: physical well-being, social/family well-being, relationship with physician, emotional well-being, and functional well-being. Scoring the FACT-G is performed through a simple sum of item scores. Each subscale is scored, and a total score for the FACT-G is obtained by adding each of the subscale scores. Higher scores for the scales and subscales indicate better quality of life in cancer patients.
Hospital Anxiety and Depression Scale | 36 months
  The Hospital Anxiety and Depression Scale (HADS), has been developed to identify caseness (possible and probable) of anxiety disorders and depression among patients in non-psychiatric hospital clinics. Concretely, it is subdivided into an Anxiety subscale (HADS-A) and a Depression subscale (HADS-D) both containing seven intermingled items. A score ≤7 corresponds to "no depression or anxiety," a score of 8-10 is a minor depression/anxiety, a score of 11-15 a moderate depression/anxiety and a score ≥16 is defined as severe depression/anxiety
Questionnaire on Distress in Cancer Patients Short-From-QSC-R10 (FBK-R10) | 36 months
  The "Questionnaire on Distress in Cancer Patients Short-From-QSC-R10" (FBK-R10) is a short questionnaire designed to measure psychological distress and burden of cancer patient. It is particularly focused on emotional distress of oncological patients. It comprises ten individual questions from the five areas: psychosomatic distress, anxiety, restrictions in everyday life, social distress and information deficit. In relation to each individual question, the patient states whether the situation applies to them and, if it does, the extent to which they feel burdened by it (rating scale from 0-5). The FBK-R10 is evaluated by summing up the indicated load strengths of the individual questions, with a possible score between 0 and 50. A Score > 14 points means positive screening for psychosocial distress.
Multidimensional Fatigue Inventory | 36 months
  The Multidimensional Fatigue Inventory (MFI) is a 20-item scale designed to assess the severity of fatigue experienced by cancer patients, as well as its impact on their ability to function33. It is designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. It can be administered in a clinical setting as part of patient screening processes and may also be useful for clinical trials. As a short scale that can be rapidly administered and easily understood, the MFI is designed to be well tolerated by patients suffering even the most severe degrees of fatigue.
Scored Patient-Generated Subjective Global Assessment | 36 months
  The Patient-Generated Subjective Global Assessment (PG-SGA) is a patient reported instrument for assessment of nutrition status in patients with cancer, as many patients have nutritional issues during or after competing their treatment regime34. It has been well characterized in patients undergoing chemo- and radiation therapy.

SECONDARY OUTCOMES:
Physiological Effects of Training | 36 months
  Physical outcomes evaluating performance will be assessed at the beginning of the 12-weeks program and immediately after completion of the program.
  Test 1: Sit-and-stand test
  The 60 Seconds Sit-to-Stand Test investigates the ability to stand up from a sitting position. The test typically assesses the maximum number of times a subject can stand up and sit down on a regular chair in each period, usually 60 Seconds.
  Test 2: Body Composition
  Body composition will be assessed by bioimpedance analysis (BIA), an electrical method of assessing human body composition with the potential of quantifying total body water, fluid volumes, body cell mass, and fat-free body mass.
  Test 3: Hand Grip Strength The Hand Grip strength will be assessed using a handgrip dynamometer. It measures the maximum isometric strength of the hand and forearm muscles, and research has shown that it may have use as a prognostic indicator for health outcomes, including cognition, mobility, functional status.
Patient Satisfaction Questionnaire | 36 months
  Patients will be asked to complete an in-depth questionnaire including closed and open-ended questions about their experience of the program to assess patient satisfaction at the end of the 12-weeks program.
6 Months Follow-Up Questionnaire | 36 months
  6 months after completion of the 12-weeks program, patients will be asked to complete an in-depth questionnaire including closed and open-ended questions about their current situation, including well-being and current participation in physical activities.
Collection of Socio-Economical Data over 12 Months after completion of the program | 36 months
  Patients socio-economical, demographic and health data are routinely collected. We will prospectively analyse patients' health data up to 12 months after completion of the program to defer health economics parameters that might help improve guidelines for physical activity in cancer patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Luzerner Kantonsspital, Lucerne, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No